CLINICAL TRIAL: NCT05633004
Title: Assessment of the Vivio System for the Non-Invasive Estimation of Left Ventricular Diastolic Pressure (LVDP) as an Aid in the Diagnosis of Heart Failure
Brief Title: Avicena LVDP Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicena LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-0001
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Vivio — Non-invasive estimation of Left-Ventricular End Diastolic Pressure (LVEDP)

SUMMARY:
The purpose of the study is to determine the relationship between non-invasive measurement of left ventricular diastolic pressure (LVDP) using the Vivio System, compared with invasively measured LVDP via direct measurement during left heart catheterization.

DETAILED DESCRIPTION:
Prospective study to document the utility of Vivio in quantifying LVDP, using directly measured LVDP collected during left heart catheterization as the comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects >21 years of age.
2. Referred for non-emergent left heart catheterization inclusive of direct measurement of LVDP as part of routine clinical management, to be performed from a femoral or radial access site.
3. Willing and able to participate in all study evaluations and allow access to medical records, including medical testing records.
4. Ability to understand and sign informed consent or have a legally authorized representative to provide informed consent on behalf of the subject.

Exclusion Criteria:

1. Acute coronary syndrome, or documented MI within a week of scheduled catheterization, cardiogenic shock, or the need for intravenous inotropic or mechanical circulatory support.
2. Carotid pulse is not palpable by a trained study researcher.
3. History of carotid sinus hypersensitivity (fainting in response to minimal touching or positioning of the neck).
4. History of significant or symptomatic carotid artery disease, including TIA, ultrasound evidence of >60% carotid stenosis, or at the discretion of the investigator; history of carotid artery stenting or surgery.
5. Open skin lesions at the site of Vivio application / examination.
6. Contraindication to placing a catheter in the LV in the judgement of the investigator (e.g., mechanical aortic valve, left ventricular thrombus, etc.).
7. Inability to obtain brachial artery blood pressure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are the sensitivity and specificity of the Vivio Cuff System for predicting elevated versus non elevated LVEDP as compared to direct measurement of LVEDP in the combined Cath Lab and Healthy Cohorts | 1 year
  The primary endpoints are the sensitivity and specificity of the Vivio Cuff System for predicting elevated versus non elevated LVEDP as compared to direct measurement of LVEDP in the combined Cath Lab and Healthy Cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided